CLINICAL TRIAL: NCT04008602
Title: Effectiveness of Quick Icing Technique on Force of Jump: Valuation Through a Jump Platform and a Mobile Application.
Brief Title: Effectiveness of Quick Icing (QI) Technique on Strenght of Jump.
Acronym: QIJ
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: Quiropraxia y Equilibrio (Other)
Responsible Party: Principal Investigator, Hernán Andrés de la Barra Ortiz, Investigator and Clinical Professor, Quiropraxia y Equilibrio
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 27062019
Record Dates: First submitted 2019-06-30; First posted 2019-07-05 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Muscle Strength
Keywords: Cooling; Criotherapy; Strenght; Plyometric exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: Quick Icing (Active Comparator): Group receiving the application of cold on the ventral side of the thigh (bilaterally) for 30 seconds, using the technique of ice beakers dynamically.
  Interventions: Device: Quick icing
- Experimental: Prolonged Cold (Active Comparator): Group receiving the intervention of "ice bag" for a period of eight minutes n the ventral side of the thigh (bilaterally).
  Interventions: Device: Prolonged Cold
- Control: (No Intervention): Group that does not receive intervention and that will rest for ten minutes.

INTERVENTIONS:
Device: Quick icing — Brief Application of cold, for a period of up to 30 seconds on a body surface which seeks to promote the activation of the nervous system to produce increased excitability.
  Other Names: Brief cooling
  Arms: Experimental: Quick Icing
Device: Prolonged Cold — Prolonged application of cold, for at least 5 minutes or more, on a body surface that aims to reduce nervous system activation by reducing the decreased nerve conduction velocity.
  Arms: Experimental: Prolonged Cold

SUMMARY:
It is known that cryotherapy has various therapeutic applications, among which are the control of the inflammatory process, resolution of edema, analgesia and decreased spasticity. In addition, the use of cold as an agent to decrease or facilitate neuromuscular activity has been documented. The scientific information that supports the relationship of short duration cold with the improvement of the motor response is scarce and outdated. The objective of this design is to evaluate the effectiveness of rapid cooling or Quick Icing technique in the improvement of muscular performance. The foregoing would be relevant in the field of Kinesiology (Physiotherapy) because it would attribute cold properties that could influence the increase in muscle strength, favoring the performance of different therapeutic exercises, training or high performance sport, in addition to supporting the proposal of this intervention in patients with particular neurological disorders.

DETAILED DESCRIPTION:
Methodology.

1. Type of study. Experimental study, randomized clinical trial.
2. Conceptual definition of the variables.

   * Jump strength: Maximum force developed by an individual for a counter-movement jump test measured in Newtons.
   * Flight time: Maximum air suspension time when performing the counter movement jump test measured in seconds.
   * Jump height: Maximum height reached by an individual for a counter movement jump test measured in centimeters for the "My Jump 2®" application.
   * Rapid cooling (Quick Icing): Short application of cold for a time not greater than thirty seconds on a body surface, seeking to promote neuromuscular excitability.
   * Prolonged cold: Application of cold for at least five minutes or more on a body surface, seeking to decrease the VCN of the underlying muscles and skin receptors.
3. Operational definition of the variables.

   * Jumping strength: It will be obtained through the program "My Jump 2®" whose software integrates the variables of flight time and height for its determination, will be measured in Newton.
   * Time of flight: "Globus Ergo Tester ®" through a processor, which time the takeoff and landing of the individual, the processor has incorporated a formula that determines the height in meters through the following h = (t2 xg) / 8 (68).
   * Jump height: On the other hand, the "My Jump 2®" application incorporates a mathematical program that determines the jump height in centimeters.
   * Quick Icing: It will be applied through the technique of ice cups on the anterior region of both thighs in the experimental group (ANNEX 5. ICE CUPS).
   * Prolonged cold: It will be applied through the ice bag technique (Ice Bag) on the anterior region of both thighs in the control group.
4. Definition of the type of variable.

   * Jump strength: Dependent, quantitative, reason variable.
   * Jump height: Dependent, quantitative, reason variable.
   * Quick cooling (Quick Icing): Independent variable, qualitative, nominal.
   * Prolonged cold: Independent variable, qualitative, nominal.
5. Sample.

   Students of the Faculty of Rehabilitation Sciences (FCR) of careers in occupational therapy and phonoaudiology, and kinesiology from the first to third year of the Andrés Bello University (UNAB).
6. Place of investigation.

   The study will be carried out in the physiotherapy laboratory of the Faculty of Rehabilitation Sciences (FCR), building C5, laboratory 401, Campus Casona Andrés Bello University, Santiago de Chile.
7. Design

This research has the characteristics of a randomized analytical experimental design (RCT). The study will be presented to the ethics committee of the Metropolitan Health Service East (SSMO) of the city of Santiago, to ensure that the study meets the necessary ethical considerations. Once the study is approved by the committee, the investigation will begin.

The sample will be determined through an intentional selection process through a participation survey constituted by closed questions. This survey will allow the selection of potential participants according to the inclusion and exclusion criteria proposed in the research. The number of participants that will make up the sample will be taken by the convenience of the researchers.

Three stages of study conduction have been designated. Stage one, called "sampling stage", will consist in the application of the survey to the students of the different levels of the three careers of the Faculty and will last for four weeks. Then the information collected will be analyzed by making a first filter in the selection of potential participants. This filter is given by the survey questions that will reflect the inclusive and exclusive criteria. A personal contact will be made of the participants that fulfill the selection characteristics and they will be invited to be part of the study. The purpose of the investigation will be explained to the potential participants and their written consent of participation will be requested. The consent document delivered will be previously approved by the bioethics committee of the Metropolitan Health Service East (SSMO), with headquarters in the Hospital Salvador, Providencia district. Stage one will last three weeks, following the planned proposal in the Gantt letter.

Stage two of the design, called the "Evaluation stage", will last four weeks according to what is proposed in the Gantt chart. This stage will consist in carrying out the ice cube test following the established evaluation protocol. With this test it will be possible to assess whether or not there are adverse responses to cold. This will allow applying a second filter of the selectable participants and who consented to participate consensually, and who were not excluded from the selection survey. Next, an assessment of the participants' ability to perform a jump type against movement in a painless way will be made in a scenario with the same environmental conditions in which the research will be carried out (Physiotherapy laboratory of the Faculty of Rehabilitation Sciences, room 401, C5). Stage two will be an instance of second filtering of the participants' selection, in order to have the people who will finally form the working groups of the study.

Stage three, called experimentation stage, will last for eight weeks. The participants will be distributed forming three working groups, a group called rapid cooling (ER), another group called prolonged cooling (EP) and a third group called control (C). The designation for each group will be previously carried out by a simple randomization process using a table of random numbers, and will be in charge of the study director. This randomization process will try to minimize the selection bias. The principal investigator will be the only one with the numbered list of the participants of each group. From this process of randomization the division of the groups will be established; G1 (ER), G2 (EP) and G3 (C). Once the three groups have been formed, an evaluator 1 will record the demographic characteristics of each participant. This record will include data such as; age, body mass index (BMI), gender and percentage of body fat. This information will be extracted from the survey of selection of the participants that will make up the groups and measurement of body fat percentage through bioimpedance. This analysis will allow to determine the homogeneity of the groups. An evaluator 2, unaware of the groups, will perform the jump measurements (counter movement mode) using the jump platform (Globus Ergo Tester®) and the mobile application (MyJump2®) following the protocol for evaluating and recording proposed data. By means of the jump platform, the flight times of each execution will be obtained, while with the mobile program the strength of the jump and height will be determined. Before performing the jump test, a five-minute pre-heating in a cycloergometer (MONARK 915E®) at a power of 80 watts will be performed. The heating will be done in the same room where the jump platform and the mobile application will be arranged. Evaluator 2 will request three jump executions in counter-movement mode (CMJ) (pre-intervention jumps) considering 15 seconds for each execution (including verbal order and execution) and leaving a rest interval of 60 seconds between each attempt.

The variables flight time, strength and height of the jump of the three executions will be tabulated in a Microsoft Excel® program template and the best values will be marked, such as "flight time, jump force and maximum pre height". Subsequently the participants will be referred to their corresponding intervention group, that is, rapid cooling (ER), prolonged cooling (EP) or control group (C). In the laboratory there will be three work boxes, one for each intervention procedure. Interveners will only have contact with the subjects belonging to their work group, without knowing the participants of the other groups, thus ensuring blinding and avoiding intervention bias.

Each participant will be 10 minutes in their respective work box. In each box an interventor will be placed. The first minute of the contemplated time will be used for the installation of each individual, leaving the remaining 9 for the intervention. The participants will be positioned lying on a stretcher with their back inclined at 45° leaving both thighs uncovered. The subjects of the Quick Icing group (G1) will be subjected to the application of cold on the front of both thighs for 30 seconds, using the technique of ice cups dynamically. Group 1 participants must wait for eight minutes for the application after they are installed. The application will be made within the last minute before ending the 10 minutes of stay in the box. The group of prolonged cold (G2) will receive the intervention of ice bag for a period of 10 minutes after the first minute of installation, which will be applied on the anterior side of the thighs. The ice pack will weigh 700 grams. The control group (G3) will not receive any intervention and will be left to rest for 10 minutes.

After 10 minutes the individuals of each group will be driven back to the jump measurement laboratory. Evaluator 2 will again record the execution of 3 jumps following the same protocol described before the intervention. The variable flight time, strength and height of the jump of the three executions will be tabulated in a Microsoft Excel® program spreadsheet and the best post-intervention values will be marked as "flight time, strength and height maximum jump post". Based on the data obtained, that is, pre and post intervention, the variables "flight time difference, force difference and jump height" will be determined for sessions 1, 2 and 3, which will allow analyzing the changes before and after the intervention. All the described measurement will be recorded as the data obtained on day 1. Participants will be instructed to repeat the same test on two other occasions, on day 3 (session 2) and on day 7 (session 3), leaving thus an interval of two days between each measurement. For session 2 and 3, the jump test will be repeated following the same protocol described and already used on day 1 of measurement.

9. Statistic analysis.

This stage will be in charge of the principal investigator, who will be responsible for storing and organizing the data collected by the evaluators. The statistical analysis of the data will be carried out with the STATA v13.0® program. The flight time, force and height jump will be considered as primary variables of the study. On the other hand, age, sex and body mass index (BMI) will be considered as secondary variables. The Shapiro Wilk test (S-Wilk) will be applied to evaluate the statistical distribution behavior of the primary variables. and height of jump pre, post and its difference. According to their statistical behavior, averages or medians will be used to represent the data. The same statistic will be applied to the secondary variables such as age and BMI to represent them as averages or medians. The secondary sex variable will be described as a function of frequencies. To perform the intra and intergroup comparisons, the ANOVA or K-WALLIS statistics will be used depending on the statistical behavior of the variables thrown by the S-Wilk test. The analysis will also consider the differences of the values obtained for the primary variables in between sessions 1, 2 and 3 of measurement.

Evaluation protocol: Ice cube test. The ice cube test involves placing an ice cube (0 to 4 °C) on the forearm for five minutes, then removing it and waiting approximately 10 minutes for the skin to return to its normal temperature. It is considered that the test is positive when there is formation of a welt or confluent welts at the place of application. It is recommended to cover the ice cube with a plastic bag to avoid contact of the skin with water. If there is wheal formation, we proceed to produce shorter stimuli with reductions of one minute, until we find the minimum time with which the patient reacts. These new exposures should be done in different sites of the forearm, to avoid negative results by degranulation of mast cells and desensitization of the skin. If there is no wheal training at the first five-minute exposure, the exposure time is increased by one minute, usually up to ten minutes; if there is no wheal training in any of these new exposures, the test is considered negative and the patient is unlikely to experience cold hives. In the scientific literature it is considered that the ice cube test has a sensitivity of 83% and a specificity of 100%.

With the ice cube test it is posible obtain three results: a negative test, a positive test during the registration period or an atypical response. Cold urticarias with an atypical response share two common characteristics: 1) clinical history of urticaria or cold angioedema, and 2) negative ice cube test immediately (except for cold reflex urticaria).

Protocol for conducting the Test.

* Subject sitting
* Shoulder position: adducted without rotation.
* Elbow position: flexed at 90º. This will be ensured by a splint.
* Forearm position: supination.
* Place an ice cube on the ventral side of the opposite forearm for a period of 5 minutes.
* Unwanted responses are observed within 10 minutes after the test. The test will be positive if there are responses such as: hives, appearance of flictenas, cold intolerance, profuse erythema or pain.

Jump protocol and parameter registration.

* The anthropometric data of each user will be recorded: age, weight and height since these are required for the use of the MyJump2® application.
* Participants will be taught the execution of the jump-against-movement (CMJ) test.
* Participants will then undergo a previous warm-up on a cycle ergometer (MONARK 915E®) for a period of five minutes. The heating will be done with a load power of 80 watts.
* After the warm-up the subjects will go to the jump platform (Globus Ergo tester®). The subject A video camera of a mobile phone will be placed in front of the subject at 1.5 meters focusing on the feet.
* For simultaneous measurement with the MyJump2® application, the subject must jump 3 times with 1-minute rest intervals. A time of 15 seconds will be consigned for the completion of each attempt. Once the 3 jumps have been made, the subjects will be taken to the intervention boxes.
* In each of the boxes it will be designated for different groups: control, cold and long-term cold and short duration, in each box will be ten minutes.
* After the intervention, the three groups will repeat the jump test.

ELIGIBILITY:
Inclusion Criteria:

* Students of the Faculty of Rehabilitation Sciences of Andrés Bello University, belonging to Occupational Therapy, Phonoaudiology and Kinesiology careers (first to third year).
* Over 18 years.
* No musculoskeletal conditions (sprains, tears, fractures, dislocations, peripheral neuropathies and contusions) in the lower extremities in the last six months.

Exclusion Criteria:

* Presence of pain or discomfort when performing the jump test against movement of the Bosco test.
* Intolerance to the cold.
* Pathologies such as cryoglobulinemia, Raynaud's disease or paroxysmal hemoglobinuria induced by cold.
* Rheumatoid diseases such as systemic lupus erythematosus, multiple myeloma or rheumatoid arthritis.
* Adverse reactions to the ice cube test (positive test).
* Osteosynthesis materials or endoprosthesis in the lower limb.

Elimination Criteria

* No tolerance to the intervention with cold that forces to suspend the treatment.
* Non-completion of the evaluation protocol (Attendance at all scheduled sessions).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Comparing maximum jump strength changes pre and post application of cold. | Baseline and 2 hours later (1 session of treatment)
  Force evaluated through movil aplication and jump plataform.

CONTACTS AND LOCATIONS:
Overall Officials: Hernán A de la Barra Ortiz, Mg., Principal Investigator — Universidad Andrés Bello
Locations (1):
- Universidad Andrés Bello, Santiago, Las Condes, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lewis M, Clayfield J. Temperature changes following quick icing: a brief investigation. Aust J Physiother. 1981 Dec;27(6):175-8. doi: 10.1016/S0004-9514(14)60756-X. PMID 25025468
- [Background] Goff B. The application of recent advances in neurophysiology to Miss M. Rood's concept of neuromuscular facilitation. Physiotherapy. 1972 Dec 10;58(12):409-15. No abstract available. PMID 4668364
- [Background] Moseley BE, Williams E. Repair of damage; DNA in bacteria. Adv Microb Physiol. 1977;16:99-156. doi: 10.1016/s0065-2911(08)60048-x. No abstract available. PMID 343549
- [Background] Oliver RA, Johnson DJ, Wheelhouse WW, Griffin PP. Isometric muscle contraction response during recovery from reduced intramuscular temperature. Arch Phys Med Rehabil. 1979 Mar;60(3):126-9. PMID 485802
- [Background] Lee JM, Warren MP, Mason SM. Effects of ice on nerve conduction velocity. Physiotherapy. 1978 Jan;64(1):2-6. No abstract available. PMID 628689
- [Background] CLARKE RS, HELLON RF, LIND AR. Vascular reactions of the human forearm to cold. Clin Sci. 1958 Feb;17(1):165-79. No abstract available. PMID 13511729
- [Background] Belitsky RB, Odam SJ, Hubley-Kozey C. Evaluation of the effectiveness of wet ice, dry ice, and cryogenic packs in reducing skin temperature. Phys Ther. 1987 Jul;67(7):1080-4. doi: 10.1093/ptj/67.7.1080. PMID 3602101
- [Background] Chesterton LS, Foster NE, Ross L. Skin temperature response to cryotherapy. Arch Phys Med Rehabil. 2002 Apr;83(4):543-9. doi: 10.1053/apmr.2002.30926. PMID 11932859
- [Background] Otte JW, Merrick MA, Ingersoll CD, Cordova ML. Subcutaneous adipose tissue thickness alters cooling time during cryotherapy. Arch Phys Med Rehabil. 2002 Nov;83(11):1501-5. doi: 10.1053/apmr.2002.34833. PMID 12422316
- [Background] Warren TA, McCarty EC, Richardson AL, Michener T, Spindler KP. Intra-articular knee temperature changes: ice versus cryotherapy device. Am J Sports Med. 2004 Mar;32(2):441-5. doi: 10.1177/0363546503258864. PMID 14977671
- [Background] Herrera E, Sandoval MC, Camargo DM, Salvini TF. Motor and sensory nerve conduction are affected differently by ice pack, ice massage, and cold water immersion. Phys Ther. 2010 Apr;90(4):581-91. doi: 10.2522/ptj.20090131. Epub 2010 Feb 25. PMID 20185615
- [Background] Van Hooren B, Zolotarjova J. The Difference Between Countermovement and Squat Jump Performances: A Review of Underlying Mechanisms With Practical Applications. J Strength Cond Res. 2017 Jul;31(7):2011-2020. doi: 10.1519/JSC.0000000000001913. PMID 28640774
- [Background] Bobbert MF, Gerritsen KG, Litjens MC, Van Soest AJ. Why is countermovement jump height greater than squat jump height? Med Sci Sports Exerc. 1996 Nov;28(11):1402-12. doi: 10.1097/00005768-199611000-00009. PMID 8933491
- [Background] Earp JE, Joseph M, Kraemer WJ, Newton RU, Comstock BA, Fragala MS, Dunn-Lewis C, Solomon-Hill G, Penwell ZR, Powell MD, Volek JS, Denegar CR, Hakkinen K, Maresh CM. Lower-body muscle structure and its role in jump performance during squat, countermovement, and depth drop jumps. J Strength Cond Res. 2010 Mar;24(3):722-9. doi: 10.1519/JSC.0b013e3181d32c04. PMID 20195084
- [Background] Ruiz-Cardenas JD, Rodriguez-Juan JJ, Rios-Diaz J. Relationship between jumping abilities and skeletal muscle architecture of lower limbs in humans: Systematic review and meta-analysis. Hum Mov Sci. 2018 Apr;58:10-20. doi: 10.1016/j.humov.2018.01.005. Epub 2018 Jan 12. PMID 29334674
- [Background] Cooper CN, Dabbs NC, Davis J, Sauls NM. Effects of Lower-Body Muscular Fatigue on Vertical Jump and Balance Performance. J Strength Cond Res. 2020 Oct;34(10):2903-2910. doi: 10.1519/JSC.0000000000002882. PMID 30273290